CLINICAL TRIAL: NCT05770206
Title: A Multi-center, Randomized, Parallel Controlled, Double-Blinded Clinical Trial to Evaluate the Effectiveness and Safety of Hydrogen-Oxygen Generator With Nebulizer for Adjuvant Treatment of Novel Coronavirus Disease 2019 (COVID-19)
Brief Title: Hydrogen-Oxygen Generator With Nebulizer for Adjuvant Treatment of Novel Coronavirus Disease 2019 (COVID-19)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weijie Guan, Doctor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMS-H-03-105
Record Dates: First submitted 2023-02-23; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Hydrogen-oxygen Gas; AMS-H-03
Keywords: Covid19; Hydrogen-oxygen Gas; AMS-H-03
MeSH Terms: conditions — COVID-19 | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Intervention Model Description: Subjects in the test group will receive treatment by using Hydrogen-Oxygen Generator with Nebulizer (manufactured by Shanghai Asclepius Meditec Co., Ltd., flow rate: 3L/min) combined with conventional basic supportive treatment (symptomatic support treatment determined by the investigator based on the condition of the subjects); subjects in the control group will receive treatment by using Medical Molecular Sieve Oxygen Generator (manufactured by Shanghai Ouliang Medical Devices Co., Ltd., flow rate: 3L/min, provided by the sponsor) combined with conventional basic supportive treatment (same with that in the test group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental Group (Experimental): Subjects in the experimental group will receive treatment by using Hydrogen-Oxygen Generator with Nebulizer (manufactured by Shanghai Asclepius Meditec Co., Ltd., flow rate: 3L/min) combined with conventional basic supportive treatment (symptomatic support treatment determined by the investigator based on the condition of the subjects);
  Interventions: Device: Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03
- Control Group (Active Comparator): subjects in the control group will receive treatment by using Medical Molecular Sieve Oxygen Generator (manufactured by Shanghai Ouliang Medical Devices Co., Ltd., flow rate: 3L/min, provided by the sponsor) combined with conventional basic supportive treatment (same with that in the test group).
  Interventions: Device: OLO-1 Medical Molecular Sieve Oxygen Generator

INTERVENTIONS:
Device: Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03 — Subjects in the experimental group will receive treatment by using Hydrogen-Oxygen Generator with Nebulizer (manufactured by Shanghai Asclepius Meditec Co., Ltd., flow rate: 3L/min) combined with conventional basic supportive treatment (symptomatic support treatment determined by the investigator based on the condition of the subjects);
  Arms: experimental Group
Device: OLO-1 Medical Molecular Sieve Oxygen Generator — subjects in the control group will receive treatment by using Medical Molecular Sieve Oxygen Generator (manufactured by Shanghai Ouliang Medical Devices Co., Ltd., flow rate: 3L/min, provided by the sponsor) combined with conventional basic supportive treatment (same with that in the test group).
  Arms: Control Group

SUMMARY:
This is a multi-center, randomized, parallel controlled, double-blinded clinical trial to evaluate the effectiveness and safety of Hydrogen-Oxygen Generator with Nebulizer for adjuvant treatment of COVID-19 patients. The test group is expected to be superior to the control group in the primary endpoint (percentage of subjects achieving clinical recovery at Day 7 of study treatment). Subjects in the test group will receive treatment by using Hydrogen-Oxygen Generator with Nebulizer (manufactured by Shanghai Asclepius Meditec Co., Ltd., flow rate: 3L/min) combined with conventional basic supportive treatment (symptomatic support treatment determined by the investigator based on the condition of the subjects); and subjects in the control group will receive treatment by using Medical Molecular Sieve Oxygen Generator (manufactured by Shanghai Ouliang Medical Devices Co., Ltd., flow rate: 3L/min, provided by the sponsor) combined with conventional basic supportive treatment (same with that in the test group).

DETAILED DESCRIPTION:
Data of the following effectiveness and safety endpoints of subjects in the two groups will be collected and analyzed in this study, including of the primary effectiveness endpoint: percentage of subjects achieving clinical recovery at Day 7 of study treatment; and the secondary effectiveness endpoints: percentage of subjects achieving clinical recovery on Day 2, 3, 5, 10 of study treatment and that before discharge; percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more on Day 2, 3, 5, 7, 10 of study treatment and before discharge; reduction of WHO Clinical Progression Scale score on Day 2, 3, 5, 7, 10 of study treatment and before discharge; changes in COVID-19 symptom scores on Day 2, 3, 5, 7, 10 of study treatment and before discharge; total length of hospital stay; time from randomization to conversion to general COVID-19; time from randomization to conversion to mild COVID-19 disease; percentage of patients with no fever, shortness of breath and chest pain on Day 2, 3, 5, 7, 10 of study treatment and before discharge; Oxygen saturation based on finger blood samples in resting non-oxygen inhalation state; and safety evaluation variables including incidences of AEs, SAEs and device deficiencies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 18 and 75 years old (inclusive).
2. Diagnosed with mild, moderate or severe type of COVID-19 according to the criteria of Scheme for Diagnosis and Treatment of 2019 Novel Coronavirus Pneumonia (Trial Version 10).
3. Positive result for COVID-19 nucleic acid test or rapid antigen detection at screening visit;
4. Presenting with at least one respiratory symptom (e.g. dyspnoea, shortness of breath) at hospital admission.
5. Be willing to participate in this trial and provide written informed consent form.

Exclusion Criteria:

1. Subjects with critical or asymptomatic type of COVID-19;
2. Subjects with any known malignant tumor or life expectancy less than half a year.
3. Subjects who are intolerable to inhalation treatment.
4. Subjects with mental disorders or cognitive impairment who are unable to provide consent.
5. Subjects with any immunodeficiency requiring chronic treatment with any corticosteroid or other immunosuppressants.
6. Complicate with any serious cardiac, hepatic or renal disease (as indicated by aspartate aminotransferase [AST] and alanine aminotransferase [ALT] ≥ 2 × upper limit of normal [ULN], or creatinine ≥ 176.8mmol/L, or New York Heart Association (NYHA) Classification for heart failure of Class IV) or any serious primary systematic disease.
7. Subjects who are going to use any non-expectorant antioxidant drug, including large doses of vitamin C and vitamin E during the study period.
8. Subjects who are participating in any other clinical study on any investigational drug or medical device.
9. Pregnant or lactating women.
10. Subjects with any other condition judged as inappropriate to participate in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the percentage of subjects with clinical recovery on Day 7 of study treatment. | Day 7of study treatment
  continuous clinical recovery is defined as score (see Appendix 2) of COVID-19 related symptoms ≤ 1 continued for 2 consecutive days or discharge criteria is met. Time of continuous clinical recovery is defined as time (days) between the first initiation of the study treatment devices and the time when the score of relevant COVID-19 related symptoms ≤ 1 continues for 2 consecutive days or discharge criteria is met (whichever comes first).

SECONDARY OUTCOMES:
Percentage of subjects achieving clinical recovery | Day 2of study treatment
  continuous clinical recovery is defined as score (see Appendix 2) of COVID-19 related symptoms ≤ 1 continued for 2 consecutive days or discharge criteria is met. Time of continuous clinical recovery is defined as time (days) between the first initiation of the study treatment devices and the time when the score of relevant COVID-19 related symptoms ≤ 1 continues for 2 consecutive days or discharge criteria is met (whichever comes first).
Percentage of subjects achieving clinical recovery | Day 3 of study treatment
  continuous clinical recovery is defined as score (see Appendix 2) of COVID-19 related symptoms ≤ 1 continued for 2 consecutive days or discharge criteria is met. Time of continuous clinical recovery is defined as time (days) between the first initiation of the study treatment devices and the time when the score of relevant COVID-19 related symptoms ≤ 1 continues for 2 consecutive days or discharge criteria is met (whichever comes first).
Percentage of subjects achieving clinical recovery | Day 5of study treatment
  continuous clinical recovery is defined as score (see Appendix 2) of COVID-19 related symptoms ≤ 1 continued for 2 consecutive days or discharge criteria is met. Time of continuous clinical recovery is defined as time (days) between the first initiation of the study treatment devices and the time when the score of relevant COVID-19 related symptoms ≤ 1 continues for 2 consecutive days or discharge criteria is met (whichever comes first).
Percentage of subjects achieving clinical recovery | Day 10 of study treatment
  continuous clinical recovery is defined as score (see Appendix 2) of COVID-19 related symptoms ≤ 1 continued for 2 consecutive days or discharge criteria is met. Time of continuous clinical recovery is defined as time (days) between the first initiation of the study treatment devices and the time when the score of relevant COVID-19 related symptoms ≤ 1 continues for 2 consecutive days or discharge criteria is met (whichever comes first).
Percentage of subjects achieving clinical recovery | through study completion, an average of 10 days
  continuous clinical recovery is defined as score (see Appendix 2) of COVID-19 related symptoms ≤ 1 continued for 2 consecutive days or discharge criteria is met. Time of continuous clinical recovery is defined as time (days) between the first initiation of the study treatment devices and the time when the score of relevant COVID-19 related symptoms ≤ 1 continues for 2 consecutive days or discharge criteria is met (whichever comes first).
Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more | Day 2 of study treatment
  Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more
Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more | Day 3 of study treatment
  Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more
Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more | Day 5 of study treatment
  Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more
Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more | Day 7 of study treatment
  Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more
Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more | Day 10 of study treatment
  Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more
Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more | The period from the beginning of treatment in patients enrolled to the time before discharge
  Percentage of subjects whose WHO Clinical Progression Scale score decreased by 1 point or more
Point reduction of WHO Clinical Progression Scale score | Day 2 of study treatment
  Point reduction of WHO Clinical Progression Scale score
Point reduction of WHO Clinical Progression Scale score | Day 3 of study treatment
  Point reduction of WHO Clinical Progression Scale score
Point reduction of WHO Clinical Progression Scale score | Day 5 of study treatment
  Point reduction of WHO Clinical Progression Scale score
Point reduction of WHO Clinical Progression Scale score | Day 7 of study treatment
  Point reduction of WHO Clinical Progression Scale score
Point reduction of WHO Clinical Progression Scale score | Day 10 of study treatment
  Point reduction of WHO Clinical Progression Scale score
Point reduction of WHO Clinical Progression Scale score | The period from the beginning of treatment in patients enrolled to the time before discharge
  Point reduction of WHO Clinical Progression Scale score
Changes in scores of COVID-19 related symptoms | Day 2 of the study treatment
  Changes in scores of COVID-19 related symptoms
Changes in scores of COVID-19 related symptoms | Day 3 of the study treatment
  Changes in scores of COVID-19 related symptoms
Changes in scores of COVID-19 related symptoms | Day 5 of the study treatment
  Changes in scores of COVID-19 related symptoms
Changes in scores of COVID-19 related symptoms | Day 7 of the study treatment
  Changes in scores of COVID-19 related symptoms
Changes in scores of COVID-19 related symptoms | Day 10 of the study treatment
  Changes in scores of COVID-19 related symptoms
Changes in scores of COVID-19 related symptoms | The period from the beginning of treatment in patients enrolled to the time before discharge
  Changes in scores of COVID-19 related symptoms
Percentage of subjects whose COVID-19 related symptoms have recovered to normal | Day 2 of the study treatment
  Percentage of subjects whose COVID-19 related symptoms have recovered to normal
Percentage of subjects whose COVID-19 related symptoms have recovered to normal | Day 3 of the study treatment
  Percentage of subjects whose COVID-19 related symptoms have recovered to normal
Percentage of subjects whose COVID-19 related symptoms have recovered to normal | Day 5 of the study treatment
  Percentage of subjects whose COVID-19 related symptoms have recovered to normal
Percentage of subjects whose COVID-19 related symptoms have recovered to normal | Day 7 of the study treatment
  Percentage of subjects whose COVID-19 related symptoms have recovered to normal
Percentage of subjects whose COVID-19 related symptoms have recovered to normal | Day 10 of the study treatment
  Percentage of subjects whose COVID-19 related symptoms have recovered to normal
Percentage of subjects whose COVID-19 related symptoms have recovered to normal | through study completion, an average of 10 days
  Percentage of subjects whose COVID-19 related symptoms have recovered to normal
Total length of hospital stay | through study completion, an average of 14 days
  Total length of hospital stay
Time from randomization to conversion to mild type of COVID-19 | Time from randomization to conversion to mild type of COVID-19
  Time from randomization to conversion to mild type of COVID-19
Oxygen saturation in resting non-oxygen inhalation state | Day 2 of study treatment
  Oxygen saturation will be measured based on finger blood samples in resting state at 10 minutes after stopping the use of the study device for subjects in the test group and the control group
Oxygen saturation in resting non-oxygen inhalation state | Day 3 of study treatment
  Oxygen saturation will be measured based on finger blood samples in resting state at 10 minutes after stopping the use of the study device for subjects in the test group and the control group
Oxygen saturation in resting non-oxygen inhalation state | Day 5 of study treatment
  Oxygen saturation will be measured based on finger blood samples in resting state at 10 minutes after stopping the use of the study device for subjects in the test group and the control group
Oxygen saturation in resting non-oxygen inhalation state | Day 7 of study treatment
  Oxygen saturation will be measured based on finger blood samples in resting state at 10 minutes after stopping the use of the study device for subjects in the test group and the control group
Oxygen saturation in resting non-oxygen inhalation state | Day 10 of study treatment
  Oxygen saturation will be measured based on finger blood samples in resting state at 10 minutes after stopping the use of the study device for subjects in the test group and the control group
Oxygen saturation in resting non-oxygen inhalation state | through study completion, an average of 10 days
  Oxygen saturation will be measured based on finger blood samples in resting state at 10 minutes after stopping the use of the study device for subjects in the test group and the control group
CRP | Day 3 of study treatment
  C-reactive protein
CRP | Day 7 of study treatment
  C-reactive protein
CRP | Day 10 of study treatment
  C-reactive protein
CRP | through study completion, an average of 10 days
  C-reactive protein
IL-6 | Day 3 of study treatment
  IL-6
IL-6 | Day 7 of study treatment
  IL-6
IL-6 | Day 10 of study treatment
  IL-6
IL-6 | through study completion, an average of 10 days
  IL-6
ferritin | Day 3 of study treatment
  ferritin
ferritin | Day 7 of study treatment
  ferritin
ferritin | Day 10 of study treatment
  ferritin
ferritin | through study completion, an average of 10 days
  ferritin
lymphocytes | Day 3 of study treatment
  lymphocytes
lymphocytes | Day 7of study treatment
  lymphocytes
lymphocytes | Day 10 of study treatment
  lymphocytes
lymphocytes | through study completion, an average of 10 days
  lymphocytes
neutrophil to lymphocyte ratio | Day 3 of study treatment
  neutrophil to lymphocyte ratio
neutrophil to lymphocyte ratio | Day 7 of study treatment
  neutrophil to lymphocyte ratio
neutrophil to lymphocyte ratio | Day 10 of study treatment
  neutrophil to lymphocyte ratio
neutrophil to lymphocyte ratio | through study completion, an average of 10 days
  neutrophil to lymphocyte ratio
Percentage of patients with fever, shortness of breath and chest pain all disappeared | Day 2 of study treatment
  Percentage of patients with fever, shortness of breath and chest pain all disappeared
Percentage of patients with fever, shortness of breath and chest pain all disappeared | Day 3 of study treatment
  Percentage of patients with fever, shortness of breath and chest pain all disappeared
Percentage of patients with fever, shortness of breath and chest pain all disappeared | Day 5 of study treatment
  Percentage of patients with fever, shortness of breath and chest pain all disappeared
Percentage of patients with fever, shortness of breath and chest pain all disappeared | Day 7 of study treatment
  Percentage of patients with fever, shortness of breath and chest pain all disappeared
Percentage of patients with fever, shortness of breath and chest pain all disappeared | Day 10 of study treatment
  Percentage of patients with fever, shortness of breath and chest pain all disappeared
Percentage of patients with fever, shortness of breath and chest pain all disappeared | through study completion, an average of 10 days
  Percentage of patients with fever, shortness of breath and chest pain all disappeared

OTHER OUTCOMES:
Incidence of AEs/SAEs | through study completion, an average of 14 days
  Definition: An AE is defined as any untoward medical occurrence during the course of the clinical trial, whether or not related to the study device. For the definition of SAE
Incidence of Device Deficiency | through study completion, an average of 14 days
  Definition: a device deficiency is defined as any inadequacy of a medical device which may pose inappropriate risks to the health or safety of the subjects under normal use of the device during the clinical trial, including inadequate labelling, quality issue, and malfunctions, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Guan Weijie, PhD, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ksiazek TG, Erdman D, Goldsmith CS, Zaki SR, Peret T, Emery S, Tong S, Urbani C, Comer JA, Lim W, Rollin PE, Dowell SF, Ling AE, Humphrey CD, Shieh WJ, Guarner J, Paddock CD, Rota P, Fields B, DeRisi J, Yang JY, Cox N, Hughes JM, LeDuc JW, Bellini WJ, Anderson LJ; SARS Working Group. A novel coronavirus associated with severe acute respiratory syndrome. N Engl J Med. 2003 May 15;348(20):1953-66. doi: 10.1056/NEJMoa030781. Epub 2003 Apr 10. PMID 12690092
- [Background] Kuiken T, Fouchier RA, Schutten M, Rimmelzwaan GF, van Amerongen G, van Riel D, Laman JD, de Jong T, van Doornum G, Lim W, Ling AE, Chan PK, Tam JS, Zambon MC, Gopal R, Drosten C, van der Werf S, Escriou N, Manuguerra JC, Stohr K, Peiris JS, Osterhaus AD. Newly discovered coronavirus as the primary cause of severe acute respiratory syndrome. Lancet. 2003 Jul 26;362(9380):263-70. doi: 10.1016/S0140-6736(03)13967-0. PMID 12892955
- [Background] Drosten C, Gunther S, Preiser W, van der Werf S, Brodt HR, Becker S, Rabenau H, Panning M, Kolesnikova L, Fouchier RA, Berger A, Burguiere AM, Cinatl J, Eickmann M, Escriou N, Grywna K, Kramme S, Manuguerra JC, Muller S, Rickerts V, Sturmer M, Vieth S, Klenk HD, Osterhaus AD, Schmitz H, Doerr HW. Identification of a novel coronavirus in patients with severe acute respiratory syndrome. N Engl J Med. 2003 May 15;348(20):1967-76. doi: 10.1056/NEJMoa030747. Epub 2003 Apr 10. PMID 12690091
- [Background] de Groot RJ, Baker SC, Baric RS, Brown CS, Drosten C, Enjuanes L, Fouchier RA, Galiano M, Gorbalenya AE, Memish ZA, Perlman S, Poon LL, Snijder EJ, Stephens GM, Woo PC, Zaki AM, Zambon M, Ziebuhr J. Middle East respiratory syndrome coronavirus (MERS-CoV): announcement of the Coronavirus Study Group. J Virol. 2013 Jul;87(14):7790-2. doi: 10.1128/JVI.01244-13. Epub 2013 May 15. No abstract available. PMID 23678167
- [Background] Zaki AM, van Boheemen S, Bestebroer TM, Osterhaus AD, Fouchier RA. Isolation of a novel coronavirus from a man with pneumonia in Saudi Arabia. N Engl J Med. 2012 Nov 8;367(19):1814-20. doi: 10.1056/NEJMoa1211721. Epub 2012 Oct 17. PMID 23075143
- [Background] Zhou ZQ, Zhong CH, Su ZQ, Li XY, Chen Y, Chen XB, Tang CL, Zhou LQ, Li SY. Breathing Hydrogen-Oxygen Mixture Decreases Inspiratory Effort in Patients with Tracheal Stenosis. Respiration. 2019;97(1):42-51. doi: 10.1159/000492031. Epub 2018 Sep 18. PMID 30227423
- [Background] Zheng ZG, Sun WZ, Hu JY, Jie ZJ, Xu JF, Cao J, Song YL, Wang CH, Wang J, Zhao H, Guo ZL, Zhong NS. Hydrogen/oxygen therapy for the treatment of an acute exacerbation of chronic obstructive pulmonary disease: results of a multicenter, randomized, double-blind, parallel-group controlled trial. Respir Res. 2021 May 13;22(1):149. doi: 10.1186/s12931-021-01740-w. PMID 33985501
- [Background] Guan WJ, Wei CH, Chen AL, Sun XC, Guo GY, Zou X, Shi JD, Lai PZ, Zheng ZG, Zhong NS. Hydrogen/oxygen mixed gas inhalation improves disease severity and dyspnea in patients with Coronavirus disease 2019 in a recent multicenter, open-label clinical trial. J Thorac Dis. 2020 Jun;12(6):3448-3452. doi: 10.21037/jtd-2020-057. No abstract available. PMID 32642277